CLINICAL TRIAL: NCT01040780
Title: A Randomized,Double-blind,Multicenter Phase III Trial to Evaluate the Safety and Efficacy of Icotinib and Gefitinib in Advanced NSCLC Patients Previously Treated With Chemotherapy
Brief Title: Safety and Efficacy Study of Icotinb in Non-small Cell Lung Cancer (NSCLC) Patients
Acronym: ICOGEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPI-2009
Record Dates: First submitted 2009-12-27; First posted 2009-12-30 (Estimated); Results first posted 2012-05-24 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Efficacy; Safety; EGFR-TKI; phase III; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Icotinib (Experimental): 125 mg three times daily (375 mg per day) by mouth
  Interventions: Drug: Icotinib
- Gefitinib (Active Comparator): 250 mg every 24 hours by mouth
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Icotinib — 125 mg three times daily (375 mg per day) by mouth
  Other Names: BPI-2009; Conmana
  Arms: Icotinib
Drug: Gefitinib — 250 mg every 24 hours by mouth
  Other Names: ZD1839; Iressa
  Arms: Gefitinib

SUMMARY:
The purpose of this study is to determine whether Icotinib is at least non-inferior to Gefitinib in the treatment of advanced non-small cell lung cancer (NSCLC) patients after one or two chemotherapies.

DETAILED DESCRIPTION:
Lung cancer is the rapidest increased type of cancer in China with over 5 times incidence rate increase during the past 30 years . It is the leading cause of death of cancer in man and 2nd in women. With the development of gefitinib and erlotinib, EGFR-TKI (epidermal growth factor receptor -tyrosine kinase inhibitor) is the most successful novel drugs developed for the treatment of these patients in recent years, especially for NSCLC patients in Asia including China. Icotinib is a novel EGFR-TKI developed by a group of Chinese scientists and clinician. It appears to be at least as good as gefitinib in terms of efficacy and better in terms of safety in phase I/II trials. In this study, a randomized, double-blind, gefitinib as control, multi-center phase III trial was designed to evaluate the safety and efficacy of icotinib in the treatment of advanced NSCLC patients after failure of 1 or 2 chemotherapy. PFS (progress free survival) is the primary end-point with OS (overall survival), ORR (objective response), TTP (time to progress), HRQOL and safety as the secondary end-point. A total of 400 patients will be recruited. EGFR and K-ras gene mutational analysis as well as a population PK study have also been proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed NSCLC with Histology or cytology; advanced （IIIb/IV).
2. Must have received 1 or 2 chemotherapy (at least 1 is platin based)before, and prior chemotherapy must be completed at least 4 weeks before study enrollment; =.

Exclusion Criteria:

1. Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Li Zhang, M.D., Principal Investigator — Sun Yat-sen University; Fenlai Tan, M.D./Ph.D., Study Director — Zhejiang Betapharma Inc.
Locations (27):
- China (27):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Bejing Cancer Hospital, Beijing, Beijing Municipality
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Third Affiliated Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Guanghzou General Hospital of PLA, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital， Southern Medical University, Guangzhou, Guangdong
  - Sun yat-sen Univerisity Cancer Center, Guanzhou, Guangdong
  - the Second Xiangya Hospital，Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - 81 Hospital of PLA, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Command，PLA, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Ruijin Hospital，Shanghai Jiao-Tong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Changhai Hospital， Second Military Medical University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - Xijing Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] Camidge DR. Icotinib: kick-starting the Chinese anticancer drug industry. Lancet Oncol. 2013 Sep;14(10):913-4. doi: 10.1016/S1470-2045(13)70385-1. Epub 2013 Aug 13. No abstract available. PMID 23948350
- [Background] Zhao Q, Shentu J, Xu N, Zhou J, Yang G, Yao Y, Tan F, Liu D, Wang Y, Zhou J. Phase I study of icotinib hydrochloride (BPI-2009H), an oral EGFR tyrosine kinase inhibitor, in patients with advanced NSCLC and other solid tumors. Lung Cancer. 2011 Aug;73(2):195-202. doi: 10.1016/j.lungcan.2010.11.007. Epub 2010 Dec 8. PMID 21144613
- [Result] Shi Y, Zhang L, Liu X, Zhou C, Zhang L, Zhang S, Wang D, Li Q, Qin S, Hu C, Zhang Y, Chen J, Cheng Y, Feng J, Zhang H, Song Y, Wu YL, Xu N, Zhou J, Luo R, Bai C, Jin Y, Liu W, Wei Z, Tan F, Wang Y, Ding L, Dai H, Jiao S, Wang J, Liang L, Zhang W, Sun Y. Icotinib versus gefitinib in previously treated advanced non-small-cell lung cancer (ICOGEN): a randomised, double-blind phase 3 non-inferiority trial. Lancet Oncol. 2013 Sep;14(10):953-61. doi: 10.1016/S1470-2045(13)70355-3. Epub 2013 Aug 13. PMID 23948351
- [Derived] Tan F, Shen X, Wang D, Xie G, Zhang X, Ding L, Hu Y, He W, Wang Y, Wang Y. Icotinib (BPI-2009H), a novel EGFR tyrosine kinase inhibitor, displays potent efficacy in preclinical studies. Lung Cancer. 2012 May;76(2):177-82. doi: 10.1016/j.lungcan.2011.10.023. Epub 2011 Nov 22. PMID 22112293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 26 Febrary 2009 and 13 November 2010 across 27 study sites.
Groups:
- Icotinib: Icotinib 125 mg three times daily (375 mg per day) by mouth
- Gefitinib: Gefitinib 250 mg every 24 hours by mouth
Period: Overall Study
Arm/Group | Icotinib | Gefitinib
Started | 200 | 199
Completed | 199 | 196
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Icotinib | Gefitinib | Total
Number analyzed (Participants) | 200 | 199 | 399
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 164 | 159 | 323
  >=65 years | 36 | 40 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.52 (10.14) | 56.43 (9.43) | 55.98 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 85 | 167
  Male | 118 | 114 | 232
Region of Enrollment [Number; unit: participants]
  China | 200 | 199 | 399

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline.
Time Frame: 2-7 months
Population: All patients who received at least one dose of study drug with measurable disease at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Icotinib | Gefitinib
Number analyzed (Participants) | 199 | 196
months | 4.6 [3.5 to 6.3] | 3.4 [2.3 to 3.8]

2. Secondary Outcome: Overall Survival
Description: Median number of months from first study treatment until time of death
Time Frame: From first study treatment until time of death
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gefitinib: 250 mg daily by mouth
Arm/Group | Icotinib | Gefitinib
Number analyzed (Participants) | 199 | 196
months | 13.3 [11.1 to 16.2] | 13.9 [11.4 to 17.3]

3. Secondary Outcome: Best Tumor Response
Description: Change in size of tumor: Complete Response (CR) = no measurable tumor; Partial Response (PR) = 30% decrease in size of measurable tumor; Stable Disease (SD) = measurable tumor size has not changed; Progressive Disease (PD) = measurable tumor larger than at baseline
Time Frame: While receiving study treatment; assessed every 21 days until progression
Measure: Number; unit: percentage of patients
Arm/Group | Icotinib | Gefitinib
Number analyzed (Participants) | 199 | 196
percentage of patients
  Complete Response (CR) | 0.5 | 0
  Partial Response (PR) | 27.1 | 27.2
  Stable Disease (SD) | 47.7 | 47.7
  Progressive Disease (PD) | 21.1 | 20.5
  Disease Control (CR+PR+SD) | 75.4 | 74.9

4. Secondary Outcome: Time To Progression
Description: Median time until disease progression. Disease progression defined as radiological and/or symptomatic disease progression.
Time Frame: 2-7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Icotinib | Gefitinib
Number analyzed (Participants) | 199 | 196
months | 5.2 [3.6 to 6.6] | 3.7 [2.5 to 5.0]

5. Secondary Outcome: Safety and Tolerability
Description: Adverse Events (AEs) and Serious AEs (SAEs) are presented regardless of causality for patients who received at least one dose of Icotinib or Gefitinib. Events were graded by the investigator using the NCI CTCAE Scale (version 3.0) which provides a grading scale for each AE term.
  Grade 3 = Severe Grade 4 = Life-threatening or disabling
Time Frame: Assessed over two years
Measure: Number; unit: participants
Arm/Group | Icotinib | Gefitinib
Number analyzed (Participants) | 200 | 199
participants
  At least one AE | 166 | 165
  At least one ADR | 121 | 140
  At least one SAE | 13 | 15
  Grade 3 and 4 AEs | 9 | 10

ADVERSE EVENTS:
Description: Events were collected by systematic assessment
Arm/Group | Icotinib | Gefitinib
Serious Adverse Events (participants affected / at risk) | 13/200 | 15/199
Other Adverse Events (participants affected / at risk) | 166/200 | 165/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icotinib (N=200) | Gefitinib (N=199)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemorrhage (General disorders) | 1 (1) | 0 (0)
Cardio-respiratory failure (Cardiac disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 2 (2)
Hospitalization due to progression (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icotinib (N=200) | Gefitinib (N=199)
Rash (Skin and subcutaneous tissue disorders) | 81 (81) | 98 (98)
Diarrhea (Gastrointestinal disorders) | 43 (43) | 58 (58)
Pain (General disorders) | 36 (36) | 22 (22)
Aminotransferase Increased (Investigations) | 21 (21) | 26 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 22 (22)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 16 (16)
Anorexia (Gastrointestinal disorders) | 11 (11) | 14 (14)
Pyrexia (General disorders) | 6 (6) | 17 (17)
Leukopenia (Blood and lymphatic system disorders) | 9 (9) | 12 (12)
Nausea (Gastrointestinal disorders) | 8 (8) | 13 (13)
Hepatic Function Abnormal (Hepatobiliary disorders) | 10 (10) | 11 (11)
Vomiting (Gastrointestinal disorders) | 9 (9) | 12 (12)
Mucositis of oral cavity (Gastrointestinal disorders) | 10 (10) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days